CLINICAL TRIAL: NCT02784561
Title: Safety and Efficacy Study of Busulfan/FLAG Conditioning Regimen in Patients With Relapsed/Refractory Acute Leukemia Undergoing Allogeneic Peripheral Blood Stem Cell Transplantation
Brief Title: Study of Busulfan and FLAG Conditioning Regimen for Allogeneic Peripheral Blood Stem Cell Transplantation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: 309th Hospital of Chinese People's Liberation Army (Other); Beijing Naval General Hospital (Other); Space Center Hospital, Peking University (Unknown)
Responsible Party: Principal Investigator, Daihong Liu, Head of Hematology departemnt in Chinese PLA General Hospital, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 81370666-2
Record Dates: First submitted 2016-05-17; First posted 2016-05-27 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Leukemia
Keywords: allogeneic peripheral blood stem cell transplantation; conditioning regimen; acute leukemia; relapsed/refractory
MeSH Terms: conditions — Leukemia; Recurrence | interventions — Busulfan; Cytarabine; fludarabine; fludarabine phosphate; Granulocyte Colony-Stimulating Factor; Antilymphocyte Serum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Busulfan/FLAG conditioning regimen (Experimental): All recipients in this arm received the conditioning regimen consisting of Busulfan/FLAG (fludarabine, cytarabine and granulocyte colony-stimulating factor).
  The conditioning regimen for peripheral blood stem cell transplantation consisted of busulfan (3.2 mg/kg/ day intravenously [i.v.], days -10 to -8), fludarabine (30 mg/m2, day -7 to -3), cytarabine (1.6 g/m2/day, days
  -7 to -3), granulocyte colony-stimulating factor (5 ug/ kg, day -8 to -3). ATG (Thymoglobuline, rabbit) for haploidentical and matched unrelated donors transplantation recipients was used on 2.5 mg/kg/d from days -5 to -2).
  Interventions: Drug: Busulfan (Zhejiang Otsuka Pharmaceutical Co. Ltd); Drug: Cytarabine(Actavis Italy S.p.A); Drug: Fludarabine (Bayer); Drug: granulocyte colony-stimulating factor (KirinKunpeng); Drug: rabbit ATG（Sanofi/Genzyme）

INTERVENTIONS:
Drug: Busulfan (Zhejiang Otsuka Pharmaceutical Co. Ltd) — busulfan (3.2 mg/kg/day intravenously [i.v.], days -10 to -8)
  Other Names: Myleran, Busulfex
Drug: Cytarabine(Actavis Italy S.p.A) — cytarabine (1.6 g/m2/day, days -7 to -3)
  Other Names: Ara-C
Drug: Fludarabine (Bayer) — fludarabine (30 mg/m2, day -7 to -3),
  Other Names: fludarabine phosphate (Fludara)
Drug: granulocyte colony-stimulating factor (KirinKunpeng) — granulocyte colony-stimulating factor (5 ug/kg, day -8 to granulocyte recovery)
  Other Names: G-CSF（granulocyte colony-stimulating factor ）
Drug: rabbit ATG（Sanofi/Genzyme） — ATG; thymoglobuline, rabbit;2.5 mg/kg/day, days -5 to -2
  Other Names: Thymoglobuline

SUMMARY:
The purpose of this study is to determine the safety and efficacy of Busulfan/FLAG (fludarabine, cytarabine and granulocyte colony-stimulating factor) Conditioning Regimen in Patients with Relapsed/refractory Acute Leukemia undergoing allogeneic peripheral blood stem cell transplantation.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (allo-SCT) is the only way to cure relapsed/refractory acute leukemia. Busulfan/Cyclophosphamide (BuCy, Cytarabine, Busulfan, Cyclophosphamide) has been a classical conditioning regimen for allo-SCT. Substitution of Cyclophosphamide in the BuCy regimen with Fludarabine (BuF) resulted in reduced toxicity and similar efficacy. FLAG (fludarabine, cytarabine and granulocyte colony-stimulating factor) is a chemotherapy regimen that has been proved to be effective for relapsed/refractory acute leukemia as salvage therapy. To reduce the relapse and improve the survival of those patients with relapsed/refractory acute leukemia who receive allo-SCT, the novel conditioning regimen consisting of Busulfan/FLAG was developed. The combination of Bu and FLAG without interval shortens the duration of conditioning and the pneutropenic period of the patient compared with successive administration of FLAG followed with BuF. In addition, regarding the established safety and efficacy of BuF and FLAG, it is reasonable to expect similar safety and enhanced antileukemic efficacy for Bu/FLAG compared with BuF. In this study, the safety and efficacy of this regimen in patients with relapsed/refractory acute leukemia undergoing allogeneic peripheral blood stem cell transplantation was investigated.

ELIGIBILITY:
Inclusion Criteria:

* relapsed/refractory acute leukemia regardless of cytogenetics
* All patients should aged 12 to 65 years
* Have matched sibling donors, ≥8/10 HLA(human leukocyte antigen) matched unrelated donors or haploidentical donors
* Patients without any uncontrolled infections or without severe pulmonary, renal, hepatic or cardiac diseases

Exclusion Criteria:

* Patients aged less than 12 years old
* Patients with any uncontrolled infections or with severe pulmonary, renal, hepatic or cardiac diseases
* Acute myeloid leukemia patients with t (15;17)

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-07; Primary Completion 2019-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants relapse as assessed by NCCN (National Comprehensive Cancer Network )criteria | two years

SECONDARY OUTCOMES:
Rate of Complete Remission as assessed by NCCN (National Comprehensive Cancer Network )criteria | 30 days
DFS(disease-free survival ) | two years
TRM(treatment-related mortality ) | two years
Number of participants with aGVHD as assessed by acute graft versus host disease grading criteria (refer to Glucksberg criteria) | three months
Number of participants with Regimen-related adverse events as assessed by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Daihong Liu, Doctor, Study Director — Chinese PLA General Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Forman SJ, Rowe JM. The myth of the second remission of acute leukemia in the adult. Blood. 2013 Feb 14;121(7):1077-82. doi: 10.1182/blood-2012-08-234492. Epub 2012 Dec 14. PMID 23243288
- [Background] Tang W, Fan X, Wang L, Hu J. Busulfan and fludarabine conditioning regimen given at hematological nadir of cytoreduction fludarabine, cytarabine, and idarubicin chemotherapy in patients with refractory acute myeloid leukemia undergoing allogeneic stem cell transplantation: a single arm pilot consort study. Medicine (Baltimore). 2015 Apr;94(15):e706. doi: 10.1097/MD.0000000000000706. PMID 25881847
- [Background] Middeke JM, Herbst R, Parmentier S, Bug G, Hanel M, Stuhler G, Schafer-Eckart K, Rosler W, Klein S, Bethge W, Bitz U, Buttner B, Knoth H, Alakel N, Schaich M, Morgner A, Kramer M, Sockel K, von Bonin M, Stolzel F, Platzbecker U, Rollig C, Thiede C, Ehninger G, Bornhauser M, Schetelig J. Clofarabine salvage therapy before allogeneic hematopoietic stem cell transplantation in patients with relapsed or refractory AML: results of the BRIDGE trial. Leukemia. 2016 Feb;30(2):261-7. doi: 10.1038/leu.2015.226. Epub 2015 Aug 18. PMID 26283567
- [Background] Fu H, Xu L, Liu D, Zhang X, Liu K, Chen H, Wang Y, Han W, Han T, Huang X. Late-onset hemorrhagic cystitis after haploidentical hematopoietic stem cell transplantation in patients with advanced leukemia: differences in ATG dosage are key. Int J Hematol. 2013 Jul;98(1):89-95. doi: 10.1007/s12185-013-1350-8. Epub 2013 Apr 30. PMID 23632950
- [Background] Wang Y, Liu QF, Xu LP, Liu KY, Zhang XH, Ma X, Fan ZP, Wu DP, Huang XJ. Haploidentical vs identical-sibling transplant for AML in remission: a multicenter, prospective study. Blood. 2015 Jun 18;125(25):3956-62. doi: 10.1182/blood-2015-02-627786. Epub 2015 May 4. PMID 25940714
- [Background] Sun Y, Beohou E, Labopin M, Volin L, Milpied N, Yakoub-Agha I, Piemontese S, Polge E, Houhou M, Huang XJ, Mohty M, Nagler A, Gorin NC; Acute Leukemia Working Party of the EBMT. Unmanipulated haploidentical versus matched unrelated donor allogeneic stem cell transplantation in adult patients with acute myelogenous leukemia in first remission: a retrospective pair-matched comparative study of the Beijing approach with the EBMT database. Haematologica. 2016 Aug;101(8):e352-4. doi: 10.3324/haematol.2015.140509. Epub 2016 Apr 14. No abstract available. PMID 27081180
- [Background] Chang YJ, Huang XJ. Haploidentical stem cell transplantation: anti-thymocyte globulin-based experience. Semin Hematol. 2016 Apr;53(2):82-9. doi: 10.1053/j.seminhematol.2016.01.004. Epub 2016 Jan 18. PMID 27000731
- [Background] Wang Y, Wu DP, Liu QF, Qin YZ, Wang JB, Xu LP, Liu YR, Zhu HH, Chen J, Dai M, Huang XJ. In adults with t(8;21)AML, posttransplant RUNX1/RUNX1T1-based MRD monitoring, rather than c-KIT mutations, allows further risk stratification. Blood. 2014 Sep 18;124(12):1880-6. doi: 10.1182/blood-2014-03-563403. PMID 25082877